CLINICAL TRIAL: NCT05247554
Title: Randomized Controlled Trial Testing the Effect of Hydroxychloroquine Combined With Low-dose Corticosteroid Therapy in Pulmonary Sarcoidosis
Brief Title: Randomized Controlled Trial of Hydroxychloroquine Combined With Low-dose Corticosteroid in Pulmonary Sarcoidosis
Acronym: QUIDOSE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP191105; 2021-001834-20 (EudraCT Number)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Sarcoidosis; Hydroxychloroquine; Pulmonary; Quality of life; Steroids
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Hydroxychloroquine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine+low-dose prednisone (Experimental): Hydroxychloroquine, tablets, 400mg/day for 6 months combined with Prednisone, 20mg/day for 1 month, then 10mg/day for 20 weeks (ie up to M6). The cumulative doses of prednisone during the 6 months of the study will be 1820mg
  Interventions: Drug: Hydroxychloroquine + low-dose prednisone
- Medium-dose prednisone (Active Comparator): "prednisone, tablets, 40mg/day for 4 weeks, then 30mg/day for 2 weeks, then 20mg/day for 2 weeks, then 15mg/day for 2 weeks, then 10mg/day for 14 weeks (i.e. up to M6).
  The cumulative doses of prednisone during the 6 months of the study will be 2870mg "
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Hydroxychloroquine + low-dose prednisone — Hydroxychloroquine, tablets, 400mg/day for 6 months combined with Prednisone, 20mg/day for 1 month, then 10mg/day for 20 weeks (ie up to M6). The cumulative doses of prednisone during the 6 months of the study will be 1820mg
  Other Names: Experimental Arm
  Arms: Hydroxychloroquine+low-dose prednisone
Drug: Prednisone — "prednisone, tablets, 40mg/day for 4 weeks, then 30mg/day for 2 weeks, then 20mg/day for 2 weeks, then 15mg/day for 2 weeks, then 10mg/day for 14 weeks (i.e. up to 6 months ).
  The cumulative doses of prednisone during the 6 months of the study will be 2870mg "
  Other Names: Standard Arm
  Arms: Medium-dose prednisone

SUMMARY:
"The reference treatment for pulmonary sarcoidosis is prolonged systemic corticosteroid therapy, which improves dyspnea, fatigue and respiratory function. However, corticosteroid therapy doesn't improve quality of life, possibly due to its adverse effects. Furthermore, in an international survey study, the first priority in treatment outcome for sarcoidosis patient was quality of life.

Hydroxychloroquine an antimalarial drug, has been shown to be effective in cutaneous and pulmonary forms of sarcoidosis but in studies with imperfect methodology. Our hypothesis is that hydroxychloroquine associated with low-dose corticosteroids improves lung function as much as ""conventional"" medium-dose corticosteroid therapy but with fewer side effects and a better quality of life in pulmonary sarcoidosis. "

DETAILED DESCRIPTION:
"Sarcoidosis is a systemic granulomatosis of unknown etiology with almost systematic pulmonary involvement. The reference treatment for pulmonary sarcoidosis is prolonged systemic corticosteroid therapy, which improves dyspnea, fatigue and respiratory function. However, corticosteroid therapy doesn't improve quality of life, possibly due to its adverse effects, which are dose- and time-dependent, such as weight gain, diabetes, insomnia, hypertension. Furthermore, in an international survey study, the first priority in treatment outcome for sarcoidosis patient was quality of life. Recent optimizations have reduced the attack treatment duration from 3 to 1 month, but with a persistence of adverse effects appearing in the first months.

Hydroxychloroquine is an antimalarial drug, used for systemic lupus erythematosus with a very good benefit/risk ratio and low cost, but also for rheumatoid arthritis. Its anti-inflammatory effects involve inhibition of antigenic presentation, chemotaxis, phagocytosis, lymphocyte proliferation, cytokine production (e.g TNFα), or Toll-like receptors expression. These immunological mechanisms are also involved in the pathogenesis of sarcoidosis. In addition, Hydroxychloroquine decreases the risk of developing diabetes mellitus, dyslipidemia or thrombotic events. Hydroxychloroquine has been shown to be effective in cutaneous and pulmonary forms of sarcoidosis, and in hypercalcemia, but in studies with imperfect methodology. Baltzan et al. showed that a maintenance treatment of hydroxychloroquine versus placebo reduced the risk of relapse and lung function decline in pulmonary sarcoidosis. Our hypothesis is that hydroxychloroquine associated with low-dose corticosteroids improves lung function as much as ""conventional"" medium-dose corticosteroid therapy but with fewer side effects and a better quality of life in pulmonary sarcoidosis. The main objective is to demonstrate the non-inferiority of the combination of hydroxychloroquine and low-dose corticosteroids versus medium-dose corticosteroid therapy on the improvement of respiratory function at 6 months.

The secondary objectives are to (i) demonstrate the superiority of the combination of hydroxychloroquine and low-dose corticosteroids versus medium-dose corticosteroid therapy at 3, 6 months and 1 year on general quality of life, respiratory quality of life, fatigue, adverse drug event, treatment compliance and (ii) demonstrate the non-inferiority of the combination of hydroxychloroquine and low-dose corticosteroids versus medium-dose corticosteroid therapy at 3, 6 months and 1 year on : respiratory function using complementary tools, respiratory symptoms, and activity of thoracic and extra-thoracic sarcoidosis. "

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* Pulmonary sarcoidosis meeting the diagnostic criteria form ATS 2020 AJRCCM diagnostic criteria.
* Patient with radiographic stage II (mediastinal-hilar bilateral lymphadenopathy and parenchymal involvement) or III (involvement pulmonary parenchymatous) and FVC<80% and respiratory symptom(s) among the following: cough, dyspnea, chest pain).
* Effective contraception for women of childbearing ages
* Informed consent signed.
* Affiliation to the social security system

Exclusion Criteria:

* Severe impairment requiring an immediate and urgent result and/or high doses of corticosteroids (neurological, cardiac, ophthalmic (severe uveitis with ocular sequala), laryngeal, nasosinusal, renal, severe hypercalcemia)
* Cardiomyopathy with heart failure
* Presence of other conditions that may influence respiratory function: COPD, Asthma, Obesity (BMI>30) pulmonary fibrosis disease, pulmonary neoplasia;
* Contraindication to hydroxychloroquinehypersensitivity to active substances or to excipients, retinopathy or severe cataract, or unilateral blindness, QTc prolongation, exposure to known treatments to prolong QT)
* Tamoxifen use
* Renal insufficiency with clearance <60ml/min
* History of retinopathy or maculopathy
* Contraindication to corticosteroid therapy (hypersensitivity of active substancies, infections and progressive virosis, glaucoma, psychotic state not controlled by treatment, live vaccine, uncontrolled diabetes mellitus and hypertension)
* Intermittent porphyria (risk of acute porphyria crisis)
* Glucose-6-Phosphate Dehydrogenase deficiency
* Seropositivity to HIV, HBV, HCV
* Systemic corticosteroid therapy or immunosuppressive therapy for at least 7 days in the previous year;
* History of treatment with hydroxychloroquine for sarcoidosis;
* Current pregnancy,
* Breastfeeding,
* Patient unable to answer questionnaires despite the presence of a caregiver.
* Patient under trustee
* Patient under legal protection
* Participation in another therapeutic interventional trial within 6 months of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage of the predicted forced vital capacity (FVC) between inclusion and 6 months | 6 months
  "Difference in percentage of the predicted forced vital capacity (FVC) between inclusion and 6 months "

CONTACTS AND LOCATIONS:
Overall Officials: Florence JENY, MD, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX DE PARIS, Hôpital Avicenne, Service de Pneumologie; Dominique VALEYRE, MD, Study Director — ASSISTANCE PUBLIQUE HOPITAUX DE PARIS, Hôpital Avicenne, Service de Pneumologie

REFERENCES:
- [Background] Broos CE, Wapenaar M, Looman CWN, In 't Veen JCCM, van den Toorn LM, Overbeek MJ, Grootenboers MJJH, Heller R, Mostard RL, Poell LHC, Hoogsteden HC, Kool M, Wijsenbeek MS, van den Blink B. Daily home spirometry to detect early steroid treatment effects in newly treated pulmonary sarcoidosis. Eur Respir J. 2018 Jan 18;51(1):1702089. doi: 10.1183/13993003.02089-2017. Print 2018 Jan. No abstract available. PMID 29348185
- [Background] Crouser ED, Maier LA, Wilson KC, Bonham CA, Morgenthau AS, Patterson KC, Abston E, Bernstein RC, Blankstein R, Chen ES, Culver DA, Drake W, Drent M, Gerke AK, Ghobrial M, Govender P, Hamzeh N, James WE, Judson MA, Kellermeyer L, Knight S, Koth LL, Poletti V, Raman SV, Tukey MH, Westney GE, Baughman RP. Diagnosis and Detection of Sarcoidosis. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2020 Apr 15;201(8):e26-e51. doi: 10.1164/rccm.202002-0251ST. PMID 32293205
- [Background] Khan NA, Donatelli CV, Tonelli AR, Wiesen J, Ribeiro Neto ML, Sahoo D, Culver DA. Toxicity risk from glucocorticoids in sarcoidosis patients. Respir Med. 2017 Nov;132:9-14. doi: 10.1016/j.rmed.2017.09.003. Epub 2017 Sep 8. PMID 29229111
- [Background] Baughman RP, Barriuso R, Beyer K, Boyd J, Hochreiter J, Knoet C, Martone F, Quadder B, Richardson J, Spitzer G, Valeyre D, Ziosi G. Sarcoidosis: patient treatment priorities. ERJ Open Res. 2018 Dec 21;4(4):00141-2018. doi: 10.1183/23120541.00141-2018. eCollection 2018 Oct. PMID 30588477
- [Background] Ponticelli C, Moroni G. Hydroxychloroquine in systemic lupus erythematosus (SLE). Expert Opin Drug Saf. 2017 Mar;16(3):411-419. doi: 10.1080/14740338.2017.1269168. Epub 2016 Dec 14. PMID 27927040
- [Background] Baltzan M, Mehta S, Kirkham TH, Cosio MG. Randomized trial of prolonged chloroquine therapy in advanced pulmonary sarcoidosis. Am J Respir Crit Care Med. 1999 Jul;160(1):192-7. doi: 10.1164/ajrccm.160.1.9809024. PMID 10390399
- [Background] Judson MA, Baughman RP, Costabel U, Flavin S, Lo KH, Kavuru MS, Drent M; Centocor T48 Sarcoidosis Investigators. Efficacy of infliximab in extrapulmonary sarcoidosis: results from a randomised trial. Eur Respir J. 2008 Jun;31(6):1189-96. doi: 10.1183/09031936.00051907. Epub 2008 Feb 6. PMID 18256069